CLINICAL TRIAL: NCT02435745
Title: Obstructive Sleep Apnoea in Ehlers-Danlos Syndrome
Acronym: OSA in EDS
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Children's Hospital, Zurich (Other); Ehlers-Danlos Network, Switzerland (Other)
Responsible Party: Principal Investigator, Malcolm Kohler, Prof. Dr. med. Malcolm Kohler, University of Zurich
Other Study IDs: KEK-ZH-Nr. 2015-0144
Record Dates: First submitted 2015-04-27; First posted 2015-05-06 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Ehlers-Danlos Syndrome; Obstructive Sleep Apnea
Keywords: Ehlers-Danlos Syndrome; Obstructive Sleep Apnea; Prevalence; Aortic Aneurysm
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Sleep Apnea, Obstructive; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ehlers-Danlos Syndrome: Patients with the diagnosis of Ehlers-Danlos syndrome
- Controls: Patients/Subjects without the diagnosis of Ehlers-Danlos syndrome

SUMMARY:
Ehlers-Danlos Syndrome (EDS) is a clinically and genetically heterogeneous group of inherited connective tissue disorders characterized by joint hypermobility, skin hyperextensibility, and tissue fragility. EDS features such as genetically related cartilage defects, craniofacial abnormalities and increased pharyngeal collapsibility have been proposed to cause obstructive sleep apnoea (OSA). There is evidence from studies based on questionnaires that EDS patients might be more frequently affected by OSA and sleep disturbances than the general population. However, the actual prevalence of OSA in patients with EDS is unknown.

Aortic root dilation and dissection are common complications of EDS and little is known about the underlying risk factors. Preliminary evidence suggests a link with OSA but this has not yet been investigated.

The primary objective of this study is to assess the prevalence of OSA in EDS-patients (100) compared to a matched control group (100). The secondary objective of this pioneer study is to assess whether there is a relationship between OSA severity and aortic diame-ter/craniofacial abnormalities in EDS patients.

DETAILED DESCRIPTION:
Ehlers-Danlos Syndrome (EDS) is a clinically and genetically heterogeneous group of inherited connective tissue disorders characterized by joint hypermobility, skin hyperextensibility, and tissue fragility. EDS features such as genetically related cartilage defects, craniofacial abnormalities and increased pharyngeal collapsibility have been proposed to cause obstructive sleep apnoea (OSA). There is evidence from studies based on questionnaires that EDS patients might be more frequently affected by OSA and sleep disturbances than the general population. However, the actual prevalence of OSA in patients with EDS is unclear.

Aortic dilation and dissection are complications associated with EDS and little is known about the underlying risk factors. Preliminary evidence suggests a link with OSA but this has not yet been investigated.

The primary objective of this study is to assess the prevalence of OSA in EDS-patients compared to a matched control group. The secondary objective of the study is to assess whether there is a relationship between OSA severity and craniofacial phenotypes / aortic diameter in EDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Diagnosis of Ehlers-Danlos Syndrome (not for control group)

Exclusion Criteria:

* Moribund or severe disease prohibiting protocol adherence
* Continuous positive airway pressure treatment for OSA during sleep study
* Physical or intellectual impairment precluding informed consent or protocol adherence
* Pregnant patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Prospective case-control study including EDS patients and controls matched for age, gender, height and weight. The following outcomes will be assessed: 1) apnoea-hypopnoea index, 2) sleep-related questionnaires, 3) medical chart review, and 4) echocardiography
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of OSA | up to 12 months

SECONDARY OUTCOMES:
Craniofacial phenotyping | up to 12 months
Aortic diameter | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, Prof. MD, Principal Investigator — University of Zurich
Locations (1):
- Division of Pulmonology, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Gaisl T, Giunta C, Bratton DJ, Sutherland K, Schlatzer C, Sievi N, Franzen D, Cistulli PA, Rohrbach M, Kohler M. Obstructive sleep apnoea and quality of life in Ehlers-Danlos syndrome: a parallel cohort study. Thorax. 2017 Aug;72(8):729-735. doi: 10.1136/thoraxjnl-2016-209560. Epub 2017 Jan 10. PMID 28073822